CLINICAL TRIAL: NCT01804894
Title: Field Tests and Their Correlation With Injury and Performance
Brief Title: Do Common Physical Tests Predict Injury or Performance
Acronym: TEAM
Status: Completed | Type: Observational
Sponsor: High Point University (Other)
Responsible Party: Principal Investigator, Eric Hegedus, Professor and Chair, Dept of Physical Therapy, High Point University
Other Study IDs: HPU-TEAMScreen
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Lower Extremity Musculoskeletal Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- athletes with lower extremity injury: athletes who were injured during one season of play

SUMMARY:
Field tests are convenient, simple tests that serve as estimates of components of athletic performance like power speed, and agility. It is thought clinically, that those who do best at these tests will perform the best in their sport and/or be the least likely to get injured. The converse is also thought to be true. The objective of this study is to administer field tests to athletes at the beginning of each season and then follow athletes over several years, tracking their injuries and their performance statistics. In this way, the investigators can determine if the clinical supposition is true and that the results of field tests are associated with injury or performance

DETAILED DESCRIPTION:
11 physical performance tests were examined to determine their ability to predict injury

ELIGIBILITY:
Inclusion Criteria:

* age18-23
* member of the university's varsity teams

Exclusion Criteria:

* injured or recently injured prior to testing
* diagnosed current neurological issue
* recent (within 6 weeks) surgery where strenuous physical testing would be contraindicated

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: college age, varsity, division 1 athletes
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
injury | 1 year

SECONDARY OUTCOMES:
performance | 1 season

OTHER OUTCOMES:
overuse injury by area of the body | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- High Point University, High Point, North Carolina, United States

REFERENCES:
- [Background] Dallinga JM, Benjaminse A, Lemmink KA. Which screening tools can predict injury to the lower extremities in team sports?: a systematic review. Sports Med. 2012 Sep 1;42(9):791-815. doi: 10.1007/BF03262295. PMID 22909185
- [Derived] Hegedus EJ, McDonough S, Bleakley C, Baxter GD, DePew JT, Bradbury I, Cook C. Physical performance tests predict injury in National Collegiate Athletic Association athletes: a three-season prospective cohort study. Br J Sports Med. 2016 Nov;50(21):1333-1337. doi: 10.1136/bjsports-2015-094885. Epub 2016 Jan 8. PMID 26746910